CLINICAL TRIAL: NCT04621851
Title: Retro-prospective Observational Study on Risk of Progression in Chronic Phase-Chronic Myeloid Leukemia Patients Eligible for Tyrosine Kinase Inhibitor Discontinuation (TFR - PRO)
Brief Title: Retro-prospective Observational Study on Risk of Progression in CP-CML Patients Eligible for TKI Discontinuation
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: TFR-PRO
Record Dates: First submitted 2020-09-14; First posted 2020-11-09 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2023-12

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Retrospective cohort: Patients who discontinued before the opening of this study will contribute to the retrospective cohort.
- Prospective cohort: Patients who will discontinue after it will contribute to the prospective cohort.
- Retrospective/Prospective cohort: Patients who discontinued before the opening of this study but will continue their discontinuation after it, will contribute to both cohorts.

SUMMARY:
The purpose of this study is to investigate the safety profile of TKI discontinuation in clinical practice, with particular regard on the risk of progression after treatment discontinuation.

DETAILED DESCRIPTION:
This study will enroll approximately 3000 CP-CML patients that must have a history of at least 4 years of TKI treatment and at least 18 months of DMR. Events developing in patients after the end of discontinuation and TKI resumption will be considered as linked to the discontinuation if they will develop within 36 months from the end of discontinuation. This rule will apply also to subsequent TD attempts. In case of a second or subsequent discontinuation attempt after the failure of a previous one (for molecular relapse), patients must have re-achieved a DMR with TKI therapy resumption and must keep DMR for at least 18 months before another TD.

Collection of data will be retrospective and prospective, as each center will collect the data for 24 months. Patients who discontinued before the opening of this study will contribute to the retrospective cohort, while those who will discontinue after it will contribute to the prospective cohort. Patients who discontinued before the opening of this study but will continue their discontinuation after it, will contribute to both cohorts. For patients prospectively recruited, monitoring of disease status will be performed to assess the maintenance of the molecular remission during the study period.

Patients with an atypical BCR-ABL1 fusion gene, which does not allow the use of Q-RT-PCR, will be monitored by qualitative PCR and will be analyzed separately. For these patients, negativity of nested qualitative RT-PCR will be considered a surrogate of DMR of patients monitored by Q-RT-PCR, while loss of negativity of first-round qualitative PCR will be considered a surrogate of loss of MMR (i.e. molecular relapse). Accordingly, for patients monitored by qualitative PCR, TKI resumption after TD will be provided in case of a new positivity of first-round PCR.

.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated IRB/IEC-approved informed consent for the prospective cohort patients.
2. Age >= 18 years.
3. Male or female patients with CML diagnosed in chronic phase (CP).
4. At least 4 years of TKI treatment.
5. At least 18 months of DMR.

Exclusion Criteria:

* Allogeneic hematopoietic stem cell transplantation.
* CML diagnosed in AP or BC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population will include all CML patients presently eligible for treatment discontinuation independently of whether they discontinued or not. For the time they did not discontinue they will contribute to the reference cohort, while after TD they will contribute data to the discontinuation cohort. In case of treatment resumption, the patient will still contribute to the discontinuation cohort for 36 months after treatment resumption, while he/she will contribute to the reference cohort thereafter, assuming a new TD did not occur.
Sampling Method: Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
The quantification of the risk of progression | 36 Month
  To quantify the risk of progression to accelerated phase (AP) or blast phase (BP), expressed as time adjusted rate (TAR), after TKI discontinuation in CML patients who undergo a first or subsequent TKI discontinuation attempt

SECONDARY OUTCOMES:
To compare the time adjusted rate (TAR) of progression from Chronic phase-Chronic Myeloid Leukemia to Accelerated phase (AP) or Blastic phase (BP) by using the percentage of blasts, promyelocytes, basophils or platelet in blood or bone marrow | 36 Month
  To compare the TAR (time adjusted rate) of progression to AP or BP that is obtained in the target population to that obtained in a similar population of patients with the same characteristics who do not discontinue TKI treatment
Progression free survival (PFS) after TKI discontinuation. | 36 Month
  PFS will be defined as time between discontinuation and progression to AP or BP.
Rate of molecular relapse (loss of MR3 or MMR) | 36 Month
  Rate of molecular relapse (loss of MR3 or MMR) at 12 and 24 months after TKI discontinuation.
Relapse free survival (RFS) after TKI discontinuation. | 36 Month
  Relapse free survival (RFS) after TKI discontinuation. RFS will be defined as time between discontinuation and loss of MMR (i.e. molecular relapse).
Percentage of relapsed patients who obtain a new deep molecular response (DMR) within 6-12 months of treatment resumption among all patients who restart TKI treatment because of a molecular relapse after TKI discontinuation. | 36 Month
  The following criteria will be used to define DMR (43):
  * MR4 = either (i) detectable disease with <0.01% BCR-ABL1IS or (ii) undetectable disease in cDNA with >10 000 ABL1 transcripts.
  * MR4.5 = either (i) detectable disease with <0.0032% BCR-ABL1IS or (ii) undetectable disease in cDNA with >32 000 ABL1 transcripts in the same volume of cDNA used to test for BCR-ABL1.
  * MR5 = either (i) detectable disease with <0.001% BCR-ABL1IS or (ii) undetectable disease in cDNA with >100 000 ABL1 transcripts in the same volume of cDNA used to test for BCR-ABL1.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Abruzzese, MD, Principal Investigator — Ospedale S. Eugenio Roma; Vincenzo Accurso, MD, Principal Investigator — A.U. Policlinico "Paolo Giaccone" Palermo; Mario Annunziata, MD, Principal Investigator — Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli" Napoli; Francesco Passamonti, MD, Principal Investigator — Ospedale di Circolo e Fondazione Macchi Varese, ASST dei Sette Laghi Varese; Massimo Bonifacio, MD, Principal Investigator — Istituti Ospitalieri di Verona- Policlinico G.B. Rossi Verona; Giovanni Caocci, MD, Principal Investigator — CTMO - Ospedale "Businco" Cagliari; Francesca Lunghi, MD, Principal Investigator — Ospedale Milano S. Raffaele Milano; Chiara Elena, MD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo di Pavia; Monica Crugnola, MD, Principal Investigator — Az Ospedaliera Universitaria Parma; Sara Galimberti, MD, Principal Investigator — Azienda Ospedaliera Pisana Pisa; Alessandra Iurlo, MD, Principal Investigator — Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano Milano; Luciano Levato, MD, Principal Investigator — Az. Ospedaliera Pugliese - Ciaccio (AOPC) Catanzaro; Maria Cristina Miggiano, MD, Principal Investigator — Azienda ULSS 8 "Berica" Ospedale San Bortolo Vicenza; Patrizia Pregno, MD, Principal Investigator — A.O. Città della Salute e della Scienza di Torino S. G.Battista Torino; Davide Rapezzi, MD, Principal Investigator — Ospedale Cuneo; Rosaria Sancetta, MD, Principal Investigator — Ospedale dell'Angelo Mestre Venezia; Fabio Stagno, MD, Principal Investigator — P.O. Gaspare Rodolico, Catania; Luigia Luciano, MD, Principal Investigator — Azienda Ospedaliera Universitaria-Università degli Studi di Napoli "Federico II"; Carmen Fava, MD, Principal Investigator — A.S.O. Ordine Mauriziano, P.O. Umberto I Torino; Philipp leCoutre, MD, Principal Investigator — Charité University of Berlin · Medical Department, Division of Oncology and Hematology; Susanne Saussele, MD, Principal Investigator — University of Mannheim; Sarit Assouline, MD, Principal Investigator — Jewish General Hospital; Alberto Álvarez-Larrán, MD, Principal Investigator — University Hospital Clínic de Barcelona
Locations (26):
- McGill University - Jewish General Hospital Division of Hematology and Department of Oncology, Montreal, Quebec, Canada
- Germany (2):
  - Charité University of Berlin - Clinic of Medicine - Hematology and Oncology, Berlin
  - University of Mannheim, Mannheim, Germania, Mannheim
- Italy (22):
  - ASST-Monza, Monza, Italy/MB
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico UOC di Ematologia, Milan, Italy/Milano
  - Universita di Tor Vergata Ospedale S. Eugenio, Rome, Italy/Rome
  - Istituto di Ematologia "Lorenzo e A. Seragnoli" Policlinico S. Orsola Malpighi,, Bologna
  - CTMO Ematologia Ospedale "Businco", Cagliari
  - Università di Catania Cattedra di Ematologia Ospedale "Ferrarotto", Catania
  - SOC Ematologia Az. Ospedaliera Pugliese Ciaccio (AOPC), Catanzaro
  - Ematologia Ospedale Cuneo, Cuneo
  - UO Ematologia O spedale Milano S. Raffaele, Miano
  - Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli", Napoli
  - Azienda Ospedaliera Universitaria Università degli Studi di Napoli "Federico II" Facoltà di Medicina e Chirurgia, Napoli
  - U.O. di Ematologia con trapianto A.U. Policlinico "Paolo Giaccone", Palermo
  - Unità operativa Ematologia e CTMO Az Ospedaliera Universitaria, Parma
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Università di Pisa Azienda Ospedaliera Pisana Divisione di Ematologia, Pisa
  - Azienda Unità Sanitaria Locale IRCCS, Reggio Emilia
  - Dipartimento di Oncologia ed Ematologia S.C. Ematologia 2 A.O. Città della Salute e della Scienza di Torino S. G.Battista, Torino
  - Struttura Complessa a Dir. Universitaria Ematologia e Terapie Cellulari A.S.O. Ordine Mauriziano, P.O. U mberto I, Torino
  - S.C. Ematologia, Ospedale di Circolo e Fondazione Macchi Varese, ASST dei Sette Laghi,, Varese
  - U.O. di Ematologia Ospedale dell'Angelo Mestre, Venezia
  - Istituti Ospitalieri di Verona Div. di Ematologia Policlinico G.B. Rossi, Verona
  - U.O. Complessa di Ematologia Azienda ULSS 8 "Berica" Ospedale San Bortolo, Vicenza
- University Hospital Clínic de Barcelona, Barcelona, Spain

DOCUMENTS (1):
  • Study Protocol (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/51/NCT04621851/Prot_000.pdf